CLINICAL TRIAL: NCT03880890
Title: (Value of Endoscopic Sphenoid Nasalization in Management of Allergic Fungal Sinusitis Involving Sphenoidal Sinus)
Brief Title: Sphenoid Nasalization in Allergic Fungal Sphenoidal Sinusitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, hoda abdelkader mohamed, ENTspechilist, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: fungal sphenoidal sinusitis
Record Dates: First submitted 2019-03-17; First posted 2019-03-19 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Fungal Sinusitis
Keywords: sphenoid nasalization

STUDY DESIGN:
Intervention Model Description: Group (A): sphenoidotomy. Group (B): Endoscopic sphenoid nasalization with posterior septectomy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sphenoidotomy (group A) (Active Comparator): sphenoidotomy opening of sphenoid sinus ostum and cleaning of the sinus
  Interventions: Procedure: sphenoidotomy versus sphenoid nasalisation
- sphenoid nasalization (group B) (Active Comparator): sphenoid nasalization in which bilateral extended sphenoidotomy, the posterior aspect of the nasal septum is resected, along with the sphenoid rostrum, the intersinus septum, and other intrasphenoid partitions, creating a common cavity with a broad drainage pathway .
  Interventions: Procedure: sphenoidotomy versus sphenoid nasalisation

INTERVENTIONS:
Procedure: sphenoidotomy versus sphenoid nasalisation — sphenoidotomy opening of sphenoid sinus ostum and cleaning of the sinus sphenoid nasalization in which bilateral extended sphenoidotomy, the posterior aspect of the nasal septum is resected, along with the sphenoid rostrum, the intersinus septum, and other intrasphenoid partitions, creating a common cavity with a broad drainage pathway .

SUMMARY:
To study the outcome of different two endoscopic sphenoid procedure for management of allergic fungal sphenoidal sinusitis : sphenoidotomy versus sphenoid nasalization with posterior septectomy .

DETAILED DESCRIPTION:
Fungal rhinosinusitis classified into invasive and noninvasive subtypes. Phenotypes of noninvasive fungal rhinosinusitis occur in immunocompetent subjects and include: local fungal colonization, fungal ball, and allergic fungal rhinosinusitis. Subtypes of invasive fungal rhinosinusitis include acute invasive fungal rhinosinusitis, chronic invasive fungal rhinosinusitis and granulomatous invasive rhinosinusitis.

The estimated incidence of sphenoid sinusitis is only 2.7% of all nasal sinus infections, also the diagnosis of sphenoid sinus fungal infection is sometimes difficult. Clinical signs are often non specific and nasal endoscopy can be strictly normal.Early diagnosis is therefore difficult and diagnosis is often delayed with headache that may sometimes persists for several years before diagnosis of the disease.

In most cases of sphenoid sinusitis, enlargement of the obstructed sinus ostium is sufficient to provide drainage of retained secretions and reestablish mucociliary clearance.According to Simmen and Jones, a type I sphenoidotomy entails identification of the ostium without further intervention; a type II sphenoidotomy entails enlargement of the ostium upward to the level of the cranial base, and inferiorly to one-half of the sinus height; and a type III sphenoidotomy involves widening the ostium to its most lateral extent.

Eloy et al in 2017 stuited that,In more extensive sphenoid sinus surgery is reserved for cases where in the disease process is extensive or previous surgery has failed. In some cases sphenoid nasalization in which bilateral extended sphenoidotomy is necessary. In this procedure, the posterior aspect of the nasal septum is resected, along with the sphenoid rostrum, the intersinus septum, and other intrasphenoid partitions, creating a common cavity with a broad drainage pathway . It also allows access to the lateral recesses of this sinus.

ELIGIBILITY:
Inclusion Criteria:

* Any age.
* Any case of allergic fungal sinusitis unilateral or bilateral involving the sphenoid sinus

Exclusion Criteria:

* Acute invasive fungal sinusitis.
* Previous Sinonasal surgery.
* Unfit patient for surgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-04 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
rate of recurrence | 6 month
  To assess the effect of nasalization of sphenoid sinus on recurrence rate of allergic fungal sinusitis Recurrence will be evaluated by clinical endoscopic evaluationof regular endoscopic examination first visit after one week,the second after 3 weeks and after 3month. CT nose and paranasal sinus will be done after 3 and 6 months.

SECONDARY OUTCOMES:
Type of caustive organism | 2weeks
  microbiological evaluation of the fungal mud will taken for culture to determine the type of the causative organism and determine if the fungal sinusitis is of invasive or non invasive type

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospital, Asyut, Egypt

REFERENCES:
- [Result] Chakrabarti A, Denning DW, Ferguson BJ, Ponikau J, Buzina W, Kita H, Marple B, Panda N, Vlaminck S, Kauffmann-Lacroix C, Das A, Singh P, Taj-Aldeen SJ, Kantarcioglu AS, Handa KK, Gupta A, Thungabathra M, Shivaprakash MR, Bal A, Fothergill A, Radotra BD. Fungal rhinosinusitis: a categorization and definitional schema addressing current controversies. Laryngoscope. 2009 Sep;119(9):1809-18. doi: 10.1002/lary.20520. PMID 19544383
- [Result] Rodrigues J, Caruthers C, Azmeh R, Dykewicz MS, Slavin RG, Knutsen AP. The spectrum of allergic fungal diseases of the upper and lower airways. Expert Rev Clin Immunol. 2016;12(5):531-50. doi: 10.1586/1744666X.2016.1142874. Epub 2016 Feb 19. PMID 26776889
- [Result] Lee TJ, Huang SF, Chang PH. Characteristics of isolated sphenoid sinus aspergilloma: report of twelve cases and literature review. Ann Otol Rhinol Laryngol. 2009 Mar;118(3):211-7. doi: 10.1177/000348940911800309. PMID 19374153
- [Result] Kwon MO, Kim KS. Headache induced by isolated sphenoid fungal sinusitis: sinus headache? J Headache Pain. 2009 Dec;10(6):473-6. doi: 10.1007/s10194-009-0153-z. Epub 2009 Sep 10. PMID 19763769
- [Result] Kieff DA, Busaba N. Treatment of isolated sphenoid sinus inflammatory disease by endoscopic sphenoidotomy without ethmoidectomy. Laryngoscope. 2002 Dec;112(12):2186-8. doi: 10.1097/00005537-200212000-00011. PMID 12461338
- [Result] Eloy JA, Marchiano E, Vazquez A. Extended Endoscopic and Open Sinus Surgery for Refractory Chronic Rhinosinusitis. Otolaryngol Clin North Am. 2017 Feb;50(1):165-182. doi: 10.1016/j.otc.2016.08.013. PMID 27888912